CLINICAL TRIAL: NCT02341781
Title: A Multicenter, Observational Study to Evaluate the Effectiveness of Lenalidomide (Revlimid®) in Subjects With Mantle Cell Lymphoma Who Have Relapsed or Progressed After Treatment With Ibrutinib or Are Refractory or Intolerant to Ibrutinib.
Brief Title: Observational Study of Lenalidomide in Subjects With Mantle Cell Lymphoma Who Failed Ibrutinib Treatment
Acronym: MCL-004
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: CC-5013-MCL-004
Record Dates: First submitted 2015-01-14; First posted 2015-01-19 (Estimated); Last update posted 2017-01-26 (Estimated); Status verified 2017-01

CONDITIONS: Lymphoma, Mantle-Cell
Keywords: MANTLE CELL LYMPHOMA; Multicenter; Observational; Lenalidomide (Revlimid®); Relapsed or progressed; Ibrutinib
MeSH Terms: conditions — Lymphoma, Mantle-Cell; Recurrence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Relapsed,Progressed,Refractory or Intolerant to ibrutinib: MCL subjects who received lenalidomide after having relapsed or progressed on ibrutinib treatment or were refractory or intolerant to ibrutinib treatment

SUMMARY:
The objective of this study is to determine the effectiveness of lenalidomide in subjects with relapsed or refractory Mantle Cell Lymphoma (MCL) following ibrutinib treatment. MCL subjects who require treatment after receiving ibrutinib therapy are considered a population with high unmet medical need. It is therefore of benefit to have data on the outcomes of treatment options available in this patient population.

An observational study design was chosen to collect the clinical data already existing or being collected for MCL subjects being treated with lenalidomide.

MCL subjects who received lenalidomide either as monotherapy or as combination treatment after having relapsed or progressed on ibrutinib treatment or were refractory or intolerant to ibrutinib treatment are eligible for the study. Lenalidomide does not need to be the next subsequent treatment after ibrutinib.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign an informed consent document (ICD), if applicable, prior to any collection of study-related data.
2. Males or females ≥ 18 years of age at the time of signing the ICD (if informed consent is applicable)
3. Diagnosis of Mantle Cell Lymphoma (MCL) as assessed by the investigator. A copy of a pathology report establishing the diagnosis of MCL must be available
4. Must have received at least one dose of ibrutinib and must have met at least one of the following criteria:

A. Relapse: Subjects with relapse following initial response of CR to ibrutinib (or an ibrutinib-containing regimen). Subjects may have discontinued or completed ibrutinib treatment at the time of relapse, and there is no upper limit on the time between the last dose of ibrutinib to time of relapse. B. Progressive disease (PD): Subjects with PD following initial response of PR to ibrutinib (or an ibrutinib-containing regimen). Subjects may have discontinued or completed ibrutinib at the time of progression, and there is no upper limit on the time between the last dose of ibrutinib to time of progression. C. Refractoriness: Subjects with i. Best response of stable disease (SD) during treatment with ibrutinib (or an ibrutinib-containing regimen), and then subsequently had PD, or ii. Best response of PD at anytime while on ibrutinib (or an ibrutinib-containing regimen) D. Intolerance: Subjects requiring premature discontinuation of ibrutinib for reasons other than PD prior to the planned end of treatment. Potential reasons for premature discontinuation may include Adverse Event (AE) attributed to ibrutinib or inability to continue ibrutinib for other reasons. Subjects responding to ibrutinib treatment must have documented PD/relapse following discontinuation of ibrutinib. The reason for the premature discontinuation of ibrutinib will be recorded.

Exclusion Criteria:

* no exclusion criteria.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Mantle Cell Lymphoma (MCL) subjects who received lenalidomide, either as monotherapy or as combination treatment, after having relapsed or progressed on ibrutinib treatment or were refractory or intolerant to ibrutinib treatment.
  Lenalidomide does not need to be the next subsequent treatment after ibrutinib.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2015-04; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Approximately 5.7 years
  Overall Response is defined as best response of Partial Remission (PR) or Complete Remission (CR) at any time during lenalidomide treatment.

SECONDARY OUTCOMES:
Duration of response (DoR) | Approximately 5.7 years
  DoR is defined as the time from the date of the initial response of at least PR (PR or CR) to the date of progressive disease (PD) or relapse.
Adverse Events | Approximately 5.7 years
  Number of participants with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Manzke, MD, Study Director — Celgene Corporation
Locations (14):
- United States (11):
  - Mayo Clinic Scottsdale, Phoenix, Arizona
  - Innovative Clinical Research Institute, Whittier, California
  - University of Miami and Sylvester Comprehensive Cancer, Miami, Florida
  - University of Michigan Comprehensive Cancer Center Division of Hematology Oncology, Ann Arbor, Michigan
  - Columbia Comprehensive Cancer Care Clinic, Jefferson City, Missouri
  - Hackensack University Medical Center, Hackensack, New Jersey
  - Weill Cornell Medical College, New York, New York
  - Levine Cancer Institute, Charlotte, North Carolina
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Froedtert and The Medical College of Wisconsin, Milwaukee, Wisconsin
- Universitatsmedizin der Johannes Gutenberg- Universitat, Mainz, Rhineland-Palatinate, Germany
- Azienda Ospedaliero Universitaria Di Bologna - Policlinico S.Orsola Malpighi, Bologna, Emilia-Romagna, Italy
- Derriford Hospital Plymouth Oncology Center Clinical, Plymouth, Devon, United Kingdom

REFERENCES:
- [Derived] Wang M, Schuster SJ, Phillips T, Lossos IS, Goy A, Rule S, Hamadani M, Ghosh N, Reeder CB, Barnett E, Bravo MC, Martin P. Observational study of lenalidomide in patients with mantle cell lymphoma who relapsed/progressed after or were refractory/intolerant to ibrutinib (MCL-004). J Hematol Oncol. 2017 Nov 2;10(1):171. doi: 10.1186/s13045-017-0537-5. PMID 29096668